CLINICAL TRIAL: NCT05202132
Title: Pilot Study on the Accuracy of Masticatory Function Assessment to Discriminate Stage IV Periodontitis From Other Periodontitis Cases
Brief Title: Masticatory Function in the Differential Diagnosis of Stage IV Periodontitis
Status: Completed | Type: Observational
Sponsor: The European Research Group on Periodontology (ERGOPerio) (Network)
Collaborators: The University of Hong Kong (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: UW20-637
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Periodontitis
Keywords: periodontitis; Screening; diagnostic accuracy
MeSH Terms: conditions — Periodontitis | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questionnaire — A 3 item validated questionnaire assessing masticatory function
Diagnostic Test: Chewing gum test — The test is based on the ability of a subject of mixing a two colour chewing gum with 20 masticatory cycles. Mixing of the two colour chewing gum will be assessed as variance of hue in a scanned image of the flattened chewing gum. The method has been validated in independent studies.

SUMMARY:
This is a pilot diagnostic accuracy study to assess the ability to discriminate in a screening context Stage IV periodontitis from other stages of periodontitis. The index test is the assessment of masticatory dysfunction performed with a questionnaire and a chewing gum test. The reference standard is a full periodontal and functional assessment performed by a trained and calibrated specialist.

DETAILED DESCRIPTION:
This is a pilot diagnostic accuracy study. Data are derived from a cross-sectional study based on a convenience, quota sample of patients referred for dental care to the reception clinic of the Prince Philip Dental Hospital or at the Institute of Advanced Dentistry, the University of Hong Kong between October 2020 and May 2021. The study will be conducted in accordance with the current revision of the Declaration of Helsinki. Informed consent will be obtained from all participants prior to enrollment in the study. This study will follow the Standards for Reporting Diagnostic Accuracy (STARD) guidelines. To limit bias, separate calibrated examiners performed the index test (chewing gum test) and the periodontal examination used for periodontitis stage and grade diagnosis (reference standard).

To evaluate the diagnostic accuracy of masticatory function assessment for Stage IV periodontitis, logistic regression analyses will be conducted in univariate analyses and the area under the receiver operating characteristic curve (AUROC), diagnostic odds ratios (DORs), sensitivity, specificity, positive predictive values and negative predictive values will be calculated.

Multivariate logistic regression models will be applied to develop a screening algorithm for Stage IV periodontitis diagnosis including the masticatory function assessment and other candidate predictors. A backward stepwise selection method will be used (p = 0.05 for inclusion in model; p = 0.05 for removal from model). The standard nomenclature for interpreting low, moderate and high levels of accuracy will be based on sensitivity and specificity as well as the AUROC values: low level = sensitivity or specificity <60%, AUROC ≤ 0.70; moderate level = sensitivity or specificity ranging from 60% to 79%, AUROC ranging from 0.71 to 0.90; high level = sensitivity or specificity ≥ 80%, AUROC>0.90

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis subjects reporting for care at reception clinic of dental hospital

Exclusion Criteria:

* presence of temporomandibular disorders,
* subjects undergoing orthodontic treatment
* less than 12 teeth;
* subjects having received periodontal treatment in the previous 12 months;
* subjects having received antibiotic medication in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience, quota sample (equal number of subjects with stage I, II, III and IV periodontitis) of consecutive patients referred for dental care to the reception clinic of the Prince Philip Dental Hospital
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | Baseline
  Area under the receiver operating curve (AUROC)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, DMD, Principal Investigator — The European Research Group on Periodontology (ERGOPerio)
Locations (2):
- Prince Philip Dental Hospital, the Univerisity of Hong Kong, Hong Kong, China
- Faculty of Dentistry, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No